CLINICAL TRIAL: NCT01411371
Title: Catheter Ablation Versus Medical Treatment of AF in Heart Failure
Acronym: CAMTAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Professor Richard Schilling, Barts & The London NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/Q0605/47
Record Dates: First submitted 2010-07-26; First posted 2011-08-08 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2010-05

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Atrial fibrillation; Heart failure; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter Ablation (Experimental): Catheter ablation of persistent atrial fibrillation to restore normal sinus rhythm.
  Interventions: Procedure: Catheter ablation of persistent atrial fibrillation
- Medical treatment alone (Active Comparator): Patients are randomised to medical treatment alone for atrial fibrillation. Treatment will be as per current guidelines for persistent atrial fibrillation, with rate control as first line (using beta-blockers, calcium channel blockers and digoxin as indicated) and rhythm control as second line (using sotalol, dronedarone, or amiodarone as indicated). (Both groups will receive standard heart failure medication including angiotensin converting enzyme inhibitors, beta blockers, aldosterone antagonists, and diuretics as indicated).
  Interventions: Drug: Medical treatment alone

INTERVENTIONS:
Procedure: Catheter ablation of persistent atrial fibrillation — Catheter ablation of AF as described previously by our group (e.g. Hunter et al, Heart 2010).
  Arms: Catheter Ablation
Drug: Medical treatment alone — Medical treatment of persistent AF as 'normal care'. Patients are randomised to medical treatment alone for atrial fibrillation. Treatment will be as per current guidelines for persistent atrial fibrillation, with rate control as first line (using beta-blockers, calcium channel blockers and digoxin as indicated) and rhythm control as second line (using sotalol, dronedarone, or amiodarone as indicated). (Both groups will receive standard heart failure medication including angiotensin converting enzyme inhibitors, beta blockers, aldosterone antagonists, and diuretics as indicated).
  Arms: Medical treatment alone

SUMMARY:
Heart failure and atrial fibrillation (AF) often coexist, and each increases the morbidity and mortality associated with the other. The investigators hypothesized that restoration of normal sinus rhythm by catheter ablation is superior to medical treatment of AF in heart failure. This study randomizes patients with heart failure and persistent AF to medical treatment of AF or catheter ablation to restore sinus rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation
* Symptomatic heart failure

Exclusion Criteria:

* Reversible causes of heart failure
* Contraindications to catheter ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-03; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Difference in ejection fraction between groups | 6 months
  Difference in left ventricular ejection fraction between groups on echocardiography at 6 months

SECONDARY OUTCOMES:
Difference in peak VO2 between groups | 6 months
Difference in NYHA class between groups | 6 months
Difference in BNP between groups | 6 months
Difference in Quality of Life between groups | 6 months
  Using SF36 and Minnessota questionaire
Reduction in end systolic volume | 6 months compared to baseline
  Comparisson between groups of the percentage reduction in left ventricular end systolic volume at 6 months compared to baseline.
Difference in heart failure symptoms | 6 months
  Comparisson between groups in heart failure symptoms using the Minessota living with heart failure questionaire.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Schilling, MD FRCP, Principal Investigator — Professor of Cardiology, Barts & The London NHS Trust
Locations (1):
- Barts & The London NHS Trust, London, UK, United Kingdom

REFERENCES:
- [Derived] Hunter RJ, Berriman TJ, Diab I, Kamdar R, Richmond L, Baker V, Goromonzi F, Sawhney V, Duncan E, Page SP, Ullah W, Unsworth B, Mayet J, Dhinoja M, Earley MJ, Sporton S, Schilling RJ. A randomized controlled trial of catheter ablation versus medical treatment of atrial fibrillation in heart failure (the CAMTAF trial). Circ Arrhythm Electrophysiol. 2014 Feb;7(1):31-8. doi: 10.1161/CIRCEP.113.000806. Epub 2014 Jan 1. PMID 24382410